CLINICAL TRIAL: NCT00521352
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Panic Disorder (PD) With Comorbid Major Depression
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Panic Disorder With Comorbid Major Depression
Acronym: rTMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5517
Record Dates: First submitted 2007-08-23; First posted 2007-08-27 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2013-11

CONDITIONS: Panic Disorder; Major Depressive Disorder
Keywords: TMS; Dorsolateral Prefrontal Cortex
MeSH Terms: conditions — Panic Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active rTMS (Active Comparator): Active Repetitive Transcranial Magnetic Stimulation (rTMS)
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham rTMS (Sham Comparator): Sham Repetitive Transcranial Magnetic Stimulation (rTMS)
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS) — Strong electromagnetic field (~2Tesla) generated briefly (~1ms) but repetitively (1Hz) for 30min, five sessions a week for up to eight weeks.
  Other Names: Magstim, Magstim Rapid, Magstim Rapid2
  Arms: Active rTMS
Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS) — Generates a field with the same parameters as active rTMS (see active arm for parameters), however, the actual magnetic fields are blocked by an electromagnetic shield built into a sham coil. The field is impeded from stimulating the brain.
  Other Names: Magstim, Magstim Rapid, Magstim Rapid2
  Arms: Sham rTMS

SUMMARY:
This study will evaluate the efficacy of 1-Hz rTMS applied to the right Dorsolateral Prefrontal Cortex (DLPFC) in patients with Panic Disorder (PD) and comorbid Major Depressive Disorder (MDD) who have not fully responded to conventional therapies.

The investigators hypothesize that:

1. compared to sham (placebo), active rTMS will improve symptoms of PD and MDD as assessed with the Panic Disorder Severity Scale (PDSS), Hamilton Depression Rating Scale (HDRS), and Clinical Global Impression (CGI);
2. active (but not sham) rTMS will normalize levels of motor cortex excitability relative to pre-treatment baseline.

DETAILED DESCRIPTION:
This study tests the efficacy of repetitive Transcranial Magnetic Stimulation (rTMS) in the treatment of Panic Disorder (PD) with comorbid Major Depression (MDD).

Despite major advances in the treatment of PD, standard therapeutic interventions are not effective for all patients, and the most common reasons for treatment failure in PD are side effects and major depression comorbidity. rTMS is a non-invasive procedure that allows stimulation of the brain using magnetic fields. Some studies have reported that rTMS may be helpful in reducing panic and depressive symptoms. While promising, prior research has several limitations (e.g., relatively small sample sizes, relatively short durations of treatment, and lack of sham (placebo) comparison).

This study addresses the drawbacks of prior work, and will provide data that will be important in determining whether rTMS can be useful for PD patients with comorbid MDD and resistant to conventional therapies. In this trial, 20 adult outpatients with PD and comorbid MDD, that have been only partially responsive to conventional therapies, will be randomly assigned to one of two treatment groups (active low frequency (1 Hz) rTMS or sham-placebo) applied to the right Dorsolateral Prefrontal Cortex (DLPFC) daily for up to four weeks. If rTMS will be added onto ongoing pharmacotherapy, the doses must have been stable for 1 month prior to study entry. The right DLPFC was selected because it is one among several brain regions implicated in PD, and functional abnormalities in DLPFC have also been consistently replicated in MDD. Pilot work indicates that stimulation of right DLPFC with low frequency rTMS was beneficial in patients with PD and MDD. Low frequency rTMS has the added benefit of a better safety profile (i.e. low risk of seizure) compared to high frequency rTMS.

Rating scales for symptom change will be obtained at baseline, during the rTMS course, and at the end of 4 weeks of treatment. Patients who do not meet response criteria after four weeks of sham will be offered an open-label cross-over phase for an additional four weeks of daily active rTMS treatment while partial responders to either active or sham will be offered an open-label cross-over phase for an additional four weeks of daily active rTMS treatment. Patients who meet response criteria in either the randomized phase or the cross-over phase will continue routine clinical care under the supervision of their treating psychiatrist, and will be invited back for a repeat assessment at 1, 3 and 6 months to determine the persistence of benefit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of Panic Disorder and Major Depressive Disorder, as confirmed by the Structured Clinical Interview for the DSM-IV-TR (SCID)
* Residual panic attacks and MDD symptoms, defined as a total PDSS score of ≥ 20 and HDRS-17 score ≥18, despite treatment with an adequate trial of a serotonin reuptake inhibitor (SRI)
* A duration of the index episode of at least a month will be included.
* An adequate SRI trial is defined as treatment for at least 6-8 weeks on the SRI, that meets the maximum recommended dosage level for PD and MDD (fluoxetine 40-60 mg/d, sertraline 100-200 mg/d, paroxetine 40-60 mg/d, fluvoxamine 200-300 mg/d, citalopram 40-60 mg/d, escitalopram 20-30 mg/d).
* Individuals who cannot tolerate medications of class and dose at the specified duration as described above will also be included.
* Patients currently on medication must be at the same stable dose(s) for one month prior to enrollment and be willing to continue at the same dose(s) through the duration of the study.

Exclusion Criteria:

* Individuals diagnosed with bipolar disorder (lifetime), any psychotic disorder (lifetime), or an Axis II personality disorder
* A history of substance abuse or dependence within the past year (except nicotine and caffeine)
* Significant acute suicide risk will be excluded.

Other exclusion criteria include those common to every TMS protocol:

* Individuals with a clinically defined neurological disorder, with an increased risk of seizure for any reason, with a history of treatment with TMS, deep brain stimulation for any disorder will be excluded.
* Patients with cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed will be excluded.
* Current use of any investigational drug, any medications with proconvulsive action, such as bupropion, maprotiline, tricyclic antidepressant, clomipramine, classical antipsychotics, and daily use of any medications with a known inhibitory effect on cortical excitability measures (e.g., anticonvulsants, standing doses of benzodiazepines, sedative/hypnotics, and atypical antipsychotics) will not be permitted.
* If participating in psychotherapy, patients must have been in stable treatment for at least three months prior to entry into the study, with no anticipation of change in frequency therapeutic sessions, or the therapeutic focus over the duration of the TMS trial.
* Finally, current significant laboratory abnormality, known or suspected pregnancy, women who are breast-feeding or women of childbearing potential not using a medically accepted form of contraception when engaging in sexual intercourse will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Mantovani, MD, Principal Investigator — Columbia University; Sarah H Lisanby, MD, Study Chair — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Zwanzger P, Minov C, Ella R, Schule C, Baghai T, Moller HJ, Rupprecht R, Padberg F. Transcranial magnetic stimulation for panic. Am J Psychiatry. 2002 Feb;159(2):315-6. doi: 10.1176/appi.ajp.159.2.315-a. No abstract available. PMID 11823280
- [Result] Nordahl TE, Stein MB, Benkelfat C, Semple WE, Andreason P, Zametkin A, Uhde TW, Cohen RM. Regional cerebral metabolic asymmetries replicated in an independent group of patients with panic disorders. Biol Psychiatry. 1998 Nov 15;44(10):998-1006. doi: 10.1016/s0006-3223(98)00026-2. PMID 9821564
- [Result] Prasko J, Horacek J, Zalesky R, Kopecek M, Novak T, Paskova B, Skrdlantova L, Belohlavek O, Hoschl C. The change of regional brain metabolism (18FDG PET) in panic disorder during the treatment with cognitive behavioral therapy or antidepressants. Neuro Endocrinol Lett. 2004 Oct;25(5):340-8. PMID 15580167
- [Result] Pizzagalli DA, Nitschke JB, Oakes TR, Hendrick AM, Horras KA, Larson CL, Abercrombie HC, Schaefer SM, Koger JV, Benca RM, Pascual-Marqui RD, Davidson RJ. Brain electrical tomography in depression: the importance of symptom severity, anxiety, and melancholic features. Biol Psychiatry. 2002 Jul 15;52(2):73-85. doi: 10.1016/s0006-3223(02)01313-6. PMID 12113998
- [Result] Garcia-Toro M, Salva Coll J, Crespi Font M, Andres Tauler J, Aguirre Orue I, Bosch Calero C. [Panic disorder and transcranial magnetic stimulation]. Actas Esp Psiquiatr. 2002 Jul-Aug;30(4):221-4. Spanish. PMID 12217271
- [Result] Fitzgerald PB, Brown TL, Marston NA, Daskalakis ZJ, De Castella A, Kulkarni J. Transcranial magnetic stimulation in the treatment of depression: a double-blind, placebo-controlled trial. Arch Gen Psychiatry. 2003 Oct;60(10):1002-8. doi: 10.1001/archpsyc.60.9.1002. PMID 14557145
- [Result] Klein E, Kreinin I, Chistyakov A, Koren D, Mecz L, Marmur S, Ben-Shachar D, Feinsod M. Therapeutic efficacy of right prefrontal slow repetitive transcranial magnetic stimulation in major depression: a double-blind controlled study. Arch Gen Psychiatry. 1999 Apr;56(4):315-20. doi: 10.1001/archpsyc.56.4.315. PMID 10197825
- [Result] Mantovani A, Lisanby SH, Pieraccini F, Ulivelli M, Castrogiovanni P, Rossi S. Repetitive Transcranial Magnetic Stimulation (rTMS) in the treatment of panic disorder (PD) with comorbid major depression. J Affect Disord. 2007 Sep;102(1-3):277-80. doi: 10.1016/j.jad.2006.11.027. Epub 2007 Jan 9. PMID 17215046
- [Result] Mantovani A, Lisanby SH, Pieraccini F, Ulivelli M, Castrogiovanni P, Rossi S. Repetitive transcranial magnetic stimulation (rTMS) in the treatment of obsessive-compulsive disorder (OCD) and Tourette's syndrome (TS). Int J Neuropsychopharmacol. 2006 Feb;9(1):95-100. doi: 10.1017/S1461145705005729. Epub 2005 Jun 28. PMID 15982444
- [Result] Cowley DS, Ha EH, Roy-Byrne PP. Determinants of pharmacologic treatment failure in panic disorder. J Clin Psychiatry. 1997 Dec;58(12):555-61; quiz 562-3. doi: 10.4088/jcp.v58n1208. PMID 9448663
- [Derived] Mantovani A, Aly M, Dagan Y, Allart A, Lisanby SH. Randomized sham controlled trial of repetitive transcranial magnetic stimulation to the dorsolateral prefrontal cortex for the treatment of panic disorder with comorbid major depression. J Affect Disord. 2013 Jan 10;144(1-2):153-9. doi: 10.1016/j.jad.2012.05.038. Epub 2012 Aug 1. PMID 22858212
- See also: Study summary on Brain Stimulation Division web site — http://www.brainstimulation.columbia.edu/research/clinical/panic_disorder.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between January 2008 and December 2010 from the Brain Behavior Clinic and the Anxiety Disorders Clinic of New York State Psychiatric Institute/Columbia University.
Pre-assignment Details: No enrolled participant was excluded from the trial. Twenty-five patients were recruited.
Groups:
- Active: Active repetitive Transcranial Magnetic Stimulation
  Repetitive Transcranial Magnetic Stimulation (rTMS) (active) : Strong electromagnetic field (~2Tesla) generated briefly (~1ms) but repetitively (1Hz) for 30min, five sessions a week for up to eight weeks.
- Sham: Placebo repetitive Transcranial Magnetic Stimulation
  Repetitive Transcranial Magnetic Stimulation (rTMS) (sham) : Generates a field with the same parameters as active rTMS (see active arm for parameters), however, the actual magnetic fields are blocked by an electromagnetic shield built into a sham coil. The field is impeded from stimulating the brain.
Period: Overall Study
Arm/Group | Active | Sham
Started | 12 | 13
Completed | 11 | 10
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Sham | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (10) | 39.8 (13.3) | 40 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 4 | 8 | 12
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Panic Disorder Severity Scale (PDSS)
Description: The Panic Disorder Severity Scale is a questionnaire developed for measuring the severity of panic disorder symptoms.
  The PDSS consists of seven items, each rated on a 5-point scale, which ranges from 0 to 4. The items assess panic frequency, resulting distress, panic-focused anticipatory anxiety, phobic avoidance of situations and of physical sensations, impairment in occupational and social functioning. The overall assessment is made by a total score, which is calculated by summing the scores for all seven items. The total scores range from 0 to 28.
  Higher scores indicate high levels of panic symptomatology. Reduction in score from baseline indicates clinical improvement of panic symptoms.
Time Frame: 4 weeks
Measure: Number; unit: responders
Arm/Group | Active | Sham
Number analyzed (Participants) | 12 | 13
responders | 6 | 1

2. Primary Outcome: Hamilton Depression Rating Scale (HDRS), 28 Item Version
Description: The Hamilton Rating Scale for Depression (HRSD) is a multiple item questionnaire used to provide an indication of depression severity. The 28-, rather then 17- or 24-, item version was used to assess subjects in this protocol.
  28-item minimum score = 0 28-item maximum score = 84
  Higher scores indicate high levels of symptomatology. Reduction in score from baseline indicates clinical symptom improvement.
Time Frame: 4 weeks
Measure: Number; unit: responders
Arm/Group | Active | Sham
Number analyzed (Participants) | 12 | 13
responders | 3 | 1

3. Secondary Outcome: Clinical Improvement (CGI-S)
Description: Minimum CGI-S score: 1 Maximum CGI-S score: 7
  Higher scores indicate the presence of high symptom severity. Decrease in scores from baseline reflects clinical symptom improvement.
  Patients will be classified as responders with a CGI-S = 1 or 2; and partial responders CGI-S = 3.
  1. = Normal, not at all ill
  2. = Borderline mentally ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Among the most extremely ill patients
Time Frame: 4 weeks
Measure: Number; unit: responders (CGI-S = 1 or 2)
Arm/Group | Active | Sham
Number analyzed (Participants) | 12 | 13
responders (CGI-S = 1 or 2) | 6 | 1

ADVERSE EVENTS:
Arm/Group | Active | Sham
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes